CLINICAL TRIAL: NCT03914872
Title: Expanded Access Neoantigen Vaccine in Solid Tumors
Status: No longer available | Type: Expanded Access
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 19-x005
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Neoantigen DNA Vaccine — The schedule for vaccination will be weeks 1, 5, 9, 13, 17, and 21. All vaccines will occur within +/- 1 week with at least 3 weeks between vaccines.
Device: Integrated electroporation device — * Ichor Medical Systems
  * All study injections will be given intramuscularly using an integrated electroporation device
  Other Names: TDS-IM System

SUMMARY:
This is an expanded access use study. Safety data will be collected from participants.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of a solid tumor
* Pathology review demonstrates tumor cellularity of >30% in quantities sufficient to complete DNA and RNA library construction
* At least 18 years of age.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Known allergy, or history of serious adverse reaction to vaccines such as anaphylaxis, hives, or respiratory difficulty.
* Acute or chronic, clinically significant hematologic, pulmonary, cardiovascular, hepatic renal, and/or other functional abnormality that would jeopardize the health and safety of the participant as determined by the investigator based on medical history, physical examination, laboratory values, and/or diagnostic studies.
* History of syncopal or vasovagal episode as determined by medical record and history in the 12 month period prior to first vaccination administration.
* Individuals in whom a skinfold measurement of the cutaneous and subcutaneous tissue for eligible injection sites (left and right medial deltoid region) exceeds 40 mm.
* Individuals in whom the ability to observe possible local reactions at the eligible injection sites (deltoid region) is, in the opinion of the investigator, unacceptably obscured due to a physical condition or permanent body art.
* Therapeutic or traumatic metal implant in the skin or muscle of either deltoid region.
* Any chronic or active neurologic disorder, including seizures and epilepsy, excluding a single febrile seizure as a child.
* Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
* Pregnant and/or breastfeeding.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: William E Gillanders, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu